CLINICAL TRIAL: NCT01175460
Title: Phase I Study of S-1 Plus Nedaplatin With Concurrent Radiotherapy for Advanced Esophageal Cancer
Brief Title: S-1 Plus Nedaplatin With Concurrent Radiotherapy for Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, JYongling, MD, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH08
Record Dates: First submitted 2010-07-31; First posted 2010-08-04 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Esophageal Cancer
Keywords: esophageal Cancer; radiation; s-1; nedaplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiotherapy (Experimental): Thoracic radiation 60Gy over 30 fractions.Concurrently, nedaplatin was given at a fixed dose of 75 mg/m2 on Days 1, and s-1 was given on Days 1-14,repeated every 4 weeks for four cycles. The dose of s-1 was initially 60 mg/m2/day and gradually increased to determine the MTD and RD of this regimen.
  Interventions: Drug: S-1, Nedaplatin

INTERVENTIONS:
Drug: S-1, Nedaplatin — nedaplatin was given at a fixed dose of 75 mg/m2 on Days 1, and s-1 on Days 1-14, repeated every 4 weeks for four cycles. The dose of s-1 was initially 60 mg/m2/day and gradually increased to determine the MTD and RD of this regimen.

SUMMARY:
Patients with advanced esophageal cancer will receive thoracic radiation therapy 60Gy over 30 fractions,and concurrent with s-1 and nedaplatin.

DETAILED DESCRIPTION:
Purpose: To determine the maximum tolerated dose (MTD) and recommended dose (RD) of S-1 in combination with nedaplatin and thoracic radiotherapy in patients with advanced esophageal Cancer.

Methods: Thoracic radiation therapy was administered in 2Gy fractions five times weekly to a total dose of 60 Gy.Concurrently, nedaplatin was given at a fixed dose of 75 mg/m2 on Days 1, and s-1 was given on Days 1-14,repeated every 4 weeks for four cycles. The dose of s-1 was initially 60 mg/m2/day and gradually increased to determine the MTD and RD of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary squamous cell or adenocarcinoma of the esophagus
* Locoregionally advanced carcinoma of esophagus without systemic metastases
* Zubrod Performance Status 0-1;
* Patients ≥ 18 years of age;
* No hypersensitivity to E. coli -derived products;
* AGC ≥ 1500/mm3, platelets ≥ 150,000/mm3, Hgb ≥ 10 gm%, serum creatinine ≤ 1.5 mg/dl and/or calculated creatinine clearance ≥ 65 cc/min; serum calcium ≤ 11gm/dl;
* Patients with prior malignancy are eligible if curable non-melanoma skin cancer or cervical cancer in situ or disease free ≥ 5 years;
* No prior chest or upper abdomen radiotherapy; no prior systemic chemotherapy within the past 5 years; no prior esophageal or gastric surgery;
* Written informed consent.

Exclusion Criteria:

* Evidence of tracheoesophageal fistula, or invasion into the trachea or major bronchi.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior systemic chemotherapy or radiation therapy for esophageal cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of s-1 in combination with nedaplatin and thoracic radiotherapy | 3 months per patient
  the MTD will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) during treatment.

SECONDARY OUTCOMES:
Objective response rate | dependent upon results

CONTACTS AND LOCATIONS:
Overall Officials: Xianghui Du, MD, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China